CLINICAL TRIAL: NCT05398796
Title: VRC 322/DMID 21-0016: A Phase I, Dose Escalation, Open-Label Clinical Trial to Evaluate Safety, Tolerability and Immunogenicity of a Nipah Virus (NiV) mRNA Vaccine, mRNA-1215, in Healthy Adults
Brief Title: Dose Escalation, Open-Label Clinical Trial to Evaluate Safety, Tolerability and Immunogenicity of a Nipah Virus (NiV) mRNA Vaccine, mRNA-1215, in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 10000687; 000687-I
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Nipah Virus Infection
Keywords: mRNA Vaccine; Pandemic Threat; First in Human; Zoonotic Transmission
MeSH Terms: conditions — Henipavirus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): 25 mcg IM, 2 injections 4 weeks apart
  Interventions: Biological: mRNA -1215
- Group 2 (Experimental): 50 mcg IM, 2 injections 4 weeks apart
  Interventions: Biological: mRNA -1215
- Group 3 (Experimental): 100 mcg IM, 2 injections 4 weeks apart
  Interventions: Biological: mRNA -1215
- Group 4 (Experimental): 10 mcg IM, 2 injections 4 weeks apart
  Interventions: Biological: mRNA -1215

INTERVENTIONS:
Biological: mRNA -1215 — mRNA-1215 is a lipid nanoparticle dispersion containing mRNA that encodes for a secreted prefusion stabilized F component covalently linked to a G monomer (PreF/G) of a NiV Malaysian 1999 strain

SUMMARY:
Background:

Nipah virus (NiV) is transmitted from animals to humans, from humans to humans, and through contaminated food. Infected people may have a cough and trouble breathing. Some people may develop serious symptoms, such as brain infection and inflammation, that can lead to death. There are no drugs or vaccines to treat or prevent NiV infection.

Objective:

To test the safety of an experimental vaccine (mRNA-1215) for NiV. Researchers will also evaluate how participants bodies respond to the vaccine.

Eligibility:

Healthy, nonpregnant adults aged 18 to 60 years.

Design:

Participants visited the NIH clinic 13 to 15 times over 14 to 16 months.

Participants received 2 doses of the experimental vaccine at 1 month apart. The vaccine was given as a shot into the muscle of the upper arm. Participants stayed in the clinic at least 30 minutes after each vaccination.

Participants were given a diary card and a thermometer. They recorded their temperature and any other reactogenicity symptoms for 7 days after each vaccination.

During each follow-up visit, 3 to 14 tubes of blood were drawn for research.

Some participants underwent an optional procedure called apheresis. A needle is placed into a vein in each arm. Blood is removed through one needle. The blood passed through a machine that separates some of the blood cells. The rest of the blood is returned to the body through another needle.

The mRNA-1215 vaccine cannot cause NiV infection.

DETAILED DESCRIPTION:
Design:

This Phase I, dose escalation, open label clinical trial was the first study of mRNA-1215 in healthy adults to evaluate the safety, tolerability, and immunogenicity of a Nipah virus (NiV) mRNA vaccine. The hypotheses were that the vaccine would be safe, tolerable, and would elicit an immune response in healthy adults.

Study Product:

The investigational mRNA-1215 vaccine is a lipid nanoparticle dispersion containing mRNA that encodes for a secreted prefusion stabilized F component covalently linked to a G monomer (PreF/G) of a NiV Malaysian 1999 strain with a trimerization domain resulting in secretion of a trimer of heterodimers.

mRNA-1215 was co-developed by the Vaccine Research Center (VRC), National Institute of Allergy and Infectious Disease (NIAID) and ModernaTX, Inc, and manufactured by ModernaTX.

Participants:

Healthy adults, 18 to 60 years of age.

Plan:

Participants were enrolled at the NIH Clinical Center and received mRNA-1215 via intramuscular (IM) injection by needle and syringe into the deltoid muscle. A dose escalation safety evaluation occurred to ensure the safety data support proceeding to the higher dose groups. The mRNA-1215 vaccine dose for Group 4 was selected based on interim analysis of safety and immunogenicity data from Groups 1-3. Participants were evaluated for safety and immune responses through clinical observation and blood collection for safety labs at specified timepoints throughout the study. The study schema was as follows:

Study Schema

Group Participants Dose/Route Day 0 Week 4

1. 10 25 mcg IM X X
2. 10 50 mcg IM X X
3. 10 100 mcg IM X X
4. 10 10 mcg IM X X

Total **40

**Enrollment of up to 50 subjects was permitted in case additional evaluations were required for safety or immunogenicity.

Duration:

Participants were evaluated for safety and immune responses throughout the study for 52 weeks following the second vaccine dose.

ELIGIBILITY:
* INCLUSION CRITERIA:

A volunteer must meet all of the following criteria:

1. Healthy adults between the ages of 18-60 years inclusive.
2. Based on history and physical examination, in good general health and without history of any of the conditions listed in the exclusion criteria.
3. Able and willing to complete the informed consent process.
4. Available for clinic visits for 52 weeks after last product administration.
5. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
6. Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) of 18 to 35 within the 56 days prior to enrollment.

   Laboratory Criteria within 56 days before enrollment:
7. White blood cells (WBC) and differential within institutional normal range or accompanied by the site Principal Investigator (PI) or designee approval.
8. Total lymphocyte count >= 800 cells/microL.
9. Platelets = 125,000 - 500,000 cells/microL.
10. Hemoglobin within institutional normal range or accompanied by the PI or designee approval.
11. Alanine aminotransferase (ALT) <= 1.25 X institutional upper limit of normal (ULN).
12. Aspartate aminotransferase (AST) <= 1.25 X institutional ULN.
13. Alkaline phosphatase (ALP) <1.1 X institutional ULN.
14. Total bilirubin within institutional normal range or accompanied by the PI or designee approval.
15. Serum creatinine <= 1.1 X institutional ULN.
16. Negative for HIV infection by an FDA-approved method of detection

    Criteria applicable to women of childbearing potential:
17. Negative beta-human chorionic gonadotropin (Beta-HCG) pregnancy test (urine or serum) on the day of enrollment.
18. Agrees to use an effective means of birth control from at least 21 days prior to enrollment through the end of the study.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

1. Breast-feeding or planning to become pregnant during the study.
2. More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 4 weeks prior to enrollment or any within the 14 days prior to enrollment.
3. Blood products within 16 weeks prior to enrollment.
4. Any vaccine, including COVID-19 vaccines, received within 4 weeks prior to enrollment.
5. Investigational research agents within 4 weeks prior to enrollment or planning to receive investigational products while on the study
6. Current allergy treatment with allergen immunotherapy with antigen injections, unless on maintenance schedule.
7. Current anti-TB prophylaxis or therapy.
8. Known immediate hypersensitivity to any component of the study product, including polyethylene glycol (PEG).
9. Confirmed past NiV infection, prior residence in (>6 months), or planned travel for any length of time during the study to countries where NiV infection is endemic, eg. Bangladesh, India, Philippines.

   Volunteer has a history of any of the following clinically significant conditions:
10. Serious reactions to vaccines that preclude receipt of the study vaccination, including allergic reaction (anaphylaxis, urticaria or allergic reaction requiring medical intervention) to SARS-CoV-2 mRNA vaccines, as determined by the investigator
11. History of myocarditis and/or pericarditis
12. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
13. Asthma that is not well controlled
14. Diabetes mellitus (type I or II), with the exception of gestational diabetes
15. Thyroid disease that is not well controlled
16. Idiopathic urticaria within the past year
17. Autoimmune disease or immunodeficiency
18. Hypertension that is not well controlled
19. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
20. Malignancy that is active or history of malignancy that is likely to recur during the period of the study
21. Seizure disorder other than 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years.
22. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
23. Guillain-Barre Syndrome
24. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a subject s ability to give informed consent, including but not limited to clinically significant forms of: infectious diseases, drug or alcohol abuse, autoimmune diseases, psychiatric disorders, or heart disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesia K Dropulic, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared.

REFERENCES:
- [Background] Loomis RJ, Stewart-Jones GBE, Tsybovsky Y, Caringal RT, Morabito KM, McLellan JS, Chamberlain AL, Nugent ST, Hutchinson GB, Kueltzo LA, Mascola JR, Graham BS. Structure-Based Design of Nipah Virus Vaccines: A Generalizable Approach to Paramyxovirus Immunogen Development. Front Immunol. 2020 Jun 11;11:842. doi: 10.3389/fimmu.2020.00842. eCollection 2020. PMID 32595632
- [Background] Loomis RJ, DiPiazza AT, Falcone S, Ruckwardt TJ, Morabito KM, Abiona OM, Chang LA, Caringal RT, Presnyak V, Narayanan E, Tsybovsky Y, Nair D, Hutchinson GB, Stewart-Jones GBE, Kueltzo LA, Himansu S, Mascola JR, Carfi A, Graham BS. Chimeric Fusion (F) and Attachment (G) Glycoprotein Antigen Delivery by mRNA as a Candidate Nipah Vaccine. Front Immunol. 2021 Dec 8;12:772864. doi: 10.3389/fimmu.2021.772864. eCollection 2021. PMID 34956199
- [Derived] Watanabe S, Yoshikawa T, Kaku Y, Kurosu T, Fukushi S, Sugimoto S, Nishisaka Y, Fuji H, Marsh G, Maeda K, Ebihara H, Morikawa S, Shimojima M, Saijo M. Construction of a recombinant vaccine expressing Nipah virus glycoprotein using the replicative and highly attenuated vaccinia virus strain LC16m8. PLoS Negl Trop Dis. 2023 Dec 15;17(12):e0011851. doi: 10.1371/journal.pntd.0011851. eCollection 2023 Dec. PMID 38100536
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000687-I.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: mRNA-1215 25 mcg IM, 2 injections 4 weeks apart
- Group 2: mRNA-1215 50 mcg IM, 2 injections 4 weeks apart
- Group 3: mRNA-1215 100 mcg IM, 2 injections 4 weeks apart
- Group 4: mRNA-1215 10 mcg IM, 2 injections 4 weeks apart
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 10 | 10 | 10 | 10
Completed Product Administration (One (1) participant in Group 4 discontinued product administration due to elevation of total bilirubin to the Grade 3 severity level after the first dose. The IND Sponsor/PI decided not to administer the second dose of vaccine to this participant.) | 10 | 10 | 10 | 9
Completed (One (1) participant in Group 2 completed product administration but did not complete follow-up as they moved from the area.) | 10 | 9 | 10 | 10
Not Completed | 0 | 1 | 0 | 0
Not completed — Participant moved from the area | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: mRNA -1215: 25 mcg IM, 2 injections 4 weeks apart
- Group 2: mRNA -1215: 50 mcg IM, 2 injections 4 weeks apart
- Group 3: mRNA -1215: 100 mcg IM, 2 injections 4 weeks apart
- Group 4: mRNA -1215: 10 mcg IM, 2 injections 4 weeks apart
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (6.5) | 40.9 (11.1) | 36.2 (13.1) | 38.5 (11.1) | 37.4 (10.6)
Age, Customized [Count of Participants; unit: Participants]
  18-20 | 0 | 0 | 0 | 0 | 0
  21-30 | 3 | 2 | 5 | 3 | 13
  31-40 | 4 | 2 | 2 | 2 | 10
  41-50 | 3 | 4 | 0 | 5 | 12
  51-60 | 0 | 2 | 3 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 5 | 5 | 18
  Male | 8 | 4 | 5 | 5 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 10 | 9 | 10 | 9 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 1 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 2 | 5
  White | 7 | 6 | 8 | 8 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI), Mean [Mean (Standard Deviation); unit: kg/m^2] | 27.4 (2.9) | 25.4 (3.5) | 26.2 (4.1) | 27.1 (4.4) | 26.5 (3.7)
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  Under 18.5 | 0 | 0 | 0 | 0 | 0
  18.5-24.9 | 1 | 6 | 3 | 5 | 15
  25.0-29.9 | 7 | 2 | 5 | 2 | 16
  30.0-35 | 2 | 2 | 2 | 3 | 9
  Missing | 0 | 0 | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  Less than high school graduate | 0 | 0 | 0 | 0 | 0
  High school graduate/GED | 0 | 1 | 0 | 0 | 1
  College/University | 3 | 6 | 5 | 5 | 19
  Advanced degree | 7 | 3 | 5 | 5 | 20
  Not Collected | 0 | 0 | 0 | 0 | 0
NIH Employee [Count of Participants; unit: Participants]
  No | 5 | 7 | 6 | 5 | 23
  Yes | 5 | 3 | 4 | 5 | 17
  Declined to Respond | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of Product Administration
Description: Participants recorded the occurrence of solicited local symptoms on a diary card for 7 days after study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, modified from FDA Guidance - September 2007.
Time Frame: 7 days after product administration
Population: Population included all enrolled participants who received study product and provided safety data (via diary card and/or laboratory results) following vaccine administration (N=40).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 10 | 10 | 10 | 10
Participants
  Pain/Tenderness: None | 1 | 1 | 0 | 4
  Pain/Tenderness: Mild | 9 | 9 | 9 | 6
  Pain/Tenderness: Moderate | 0 | 0 | 1 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0
  Swelling: None | 10 | 10 | 9 | 10
  Swelling: Mild | 0 | 0 | 1 | 0
  Swelling: Moderate | 0 | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0 | 0
  Redness: None | 10 | 10 | 8 | 10
  Redness: Mild | 0 | 0 | 1 | 0
  Redness: Moderate | 0 | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 1 | 0
  Pruritus: None | 9 | 10 | 9 | 9
  Pruritus: Mild | 1 | 0 | 1 | 1
  Pruritus: Moderate | 0 | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0 | 0
  Axillary Lymphadenopathy Ipsilateral: None | 10 | 10 | 10 | 9
  Axillary Lymphadenopathy Ipsilateral: Mild | 0 | 0 | 0 | 1
  Axillary Lymphadenopathy Ipsilateral: Moderate | 0 | 0 | 0 | 0
  Axillary Lymphadenopathy Ipsilateral: Severe | 0 | 0 | 0 | 0
  Any Local Symptom: None | 1 | 1 | 0 | 4
  Any Local Symptom: Mild | 9 | 9 | 8 | 6
  Any Local Symptom: Moderate | 0 | 0 | 1 | 0
  Any Local Symptom: Severe | 0 | 0 | 1 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of Product Administration
Description: Participants recorded the occurrence of solicited systemic symptoms on a diary card for 7 days after study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, modified from FDA Guidance - September 2007.
Time Frame: 7 days after product administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 10 | 10 | 10 | 10
Participants
  Malaise: None | 8 | 4 | 2 | 8
  Malaise: Mild | 2 | 6 | 6 | 2
  Malaise: Moderate | 0 | 0 | 2 | 0
  Malaise: Severe | 0 | 0 | 0 | 0
  Myalgia: None | 9 | 6 | 4 | 8
  Myalgia: Mild | 1 | 4 | 5 | 2
  Myalgia: Moderate | 0 | 0 | 1 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0
  Headache: None | 6 | 6 | 4 | 9
  Headache: Mild | 4 | 3 | 6 | 1
  Headache: Moderate | 0 | 1 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0
  Chills: None | 9 | 9 | 6 | 9
  Chills: Mild | 1 | 1 | 1 | 1
  Chills: Moderate | 0 | 0 | 3 | 0
  Chills: Severe | 0 | 0 | 0 | 0
  Nausea: None | 8 | 8 | 8 | 9
  Nausea: Mild | 2 | 2 | 1 | 0
  Nausea: Moderate | 0 | 0 | 1 | 1
  Nausea: Severe | 0 | 0 | 0 | 0
  Temperature: None | 10 | 10 | 8 | 10
  Temperature: Mild | 0 | 0 | 1 | 0
  Temperature: Moderate | 0 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 1 | 0
  Joint Pain: None | 9 | 9 | 7 | 9
  Joint Pain: Mild | 1 | 1 | 3 | 1
  Joint Pain: Moderate | 0 | 0 | 0 | 0
  Joint Pain: Severe | 0 | 0 | 0 | 0
  Any Systemic Symptom: None | 6 | 4 | 2 | 7
  Any Systemic Symptom: Mild | 4 | 5 | 4 | 2
  Any Systemic Symptom: Moderate | 0 | 1 | 3 | 1
  Any Systemic Symptom: Severe | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants With Serious Adverse Events Following Product Administration
Description: SAEs were recorded from receipt of product administration through the last study visit at Week 56. The relationship between a SAE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 after product administration through Day 392, up to Week 56
Population: Population included all enrolled participants who received study product (N=40).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 10 | 10 | 10 | 10
Participants
  Related to Study Product | 0 | 0 | 0 | 0
  Unrelated to Study Product | 0 | 0 | 0 | 0
  Total Number of Participants who had SAE | 0 | 0 | 0 | 0
  Total number of Participants who did not have SAE | 10 | 10 | 10 | 10

4. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs) Following Product Administration
Description: Unsolicited AEs and attribution assessments were recorded in the study database from receipt of study product administration through the visit scheduled for 4 weeks after study product administration. At other time periods greater than 4 weeks after the study product administration, only serious AEs (SAEs reported as a separate outcome and in the AE module) and new chronic medical conditions were recorded through the last study visit. The relationship between an AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 28 days post product administration, up to Week 4
Population: Population included all enrolled participants who received study product (N=40).
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 10 | 10 | 10 | 10
participants
  Related to Study Product | 0 | 1 | 5 | 3
  Unrelated to Study Product | 5 | 5 | 7 | 7
  Total Number of Participants who had One or More Non-Serious Unsolicited AE | 5 | 5 | 7 | 8

5. Primary Outcome: Number of Participants With New Chronic Medical Conditions Following Product Administration
Description: New chronic medical conditions that required ongoing medical management were recorded from receipt of study product administration through the last expected study visit through Day 392, up to Week 56. The relationship between a new chronic medical condition and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity
Time Frame: Day 0 after product administration through Day 392, up to Week 56
Population: Population included all enrolled participants who received study product (N=40)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 10 | 10 | 10 | 10
Participants
  Related to Study Product | 0 | 0 | 0 | 0
  Unrelated to Study Product | 0 | 0 | 0 | 0
  Number of Participants With New Chronic Medical Condition | 0 | 0 | 0 | 0
  Number of Participants With No New Chronic Medical Condition | 10 | 10 | 10 | 10

6. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESI) Following Product Administration
Description: An AESI is an AE (serious or nonserious) of scientific medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the investigator to the Sponsor is required.
Time Frame: Day 0 after product administration through Day 392, up to Week 56
Population: Population included all enrolled participants who received study product (N=40)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 10 | 10 | 10 | 10
Participants
  Anaphylaxis | 0 | 0 | 0 | 0
  Myocarditis and Pericarditis | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Medically Attended Adverse Events (MAAEs) Following Product Administration
Description: MAAEs are defined as adverse events leading to hospitalization, an emergency room visit or an otherwise unscheduled visit to or from medical personnel, for any reason.
Time Frame: First vaccination to 6 months
Population: Population included all enrolled participants who received study product (N=40)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 10 | 10 | 10 | 10
Participants
  VERTEBRAL DISC HERNIATION | 1 | 0 | 0 | 0
  MUSCLE STRAIN | 0 | 1 | 0 | 0
  UPPER RESPIRATORY INFECTION | 0 | 1 | 0 | 0
  LIGAMENT TEAR | 0 | 0 | 1 | 0
  URTICARIA | 0 | 0 | 1 | 0
  PARONYCHIA | 0 | 0 | 1 | 0
  WHIPLASH | 0 | 0 | 1 | 0

8. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety Following Product Administration
Description: Abnormal lab results recorded as unsolicited adverse events (AEs) are summarized*. Safety lab parameters included pregnancy test, hematology and chemistry labs, and HIV Serology diagnostic test. Institutional lab normal ranges as well as Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials FDA Guidance, September 2007 were used.
Time Frame: Day 0 after product administration through Day 392, up to Week 56
Population: *Abnormal Laboratory Measures of Safety Following Product Administration. Participants are counted once for each category at the highest severity of AE regardless of the number of events or attribution to study vaccine.
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 10 | 10 | 10 | 10
participants
  ANEMIA : Mild | 1 | 2 | 0 | 0
  ANEMIA : Moderate | 0 | 1 | 1 | 0
  ANEMIA : Severe | 0 | 0 | 0 | 0
  ANEMIA : Total | 1 | 3 | 1 | 0
  ELEVATED AST : Mild | 1 | 0 | 0 | 0
  ELEVATED AST : Moderate | 0 | 0 | 0 | 0
  ELEVATED AST : Severe | 0 | 0 | 0 | 0
  ELEVATED AST : Total | 1 | 0 | 0 | 0
  HYPERBILIRUBINEMIA : Mild | 1 | 0 | 0 | 0
  HYPERBILIRUBINEMIA : Moderate | 0 | 0 | 0 | 0
  HYPERBILIRUBINEMIA : Severe | 0 | 0 | 0 | 1
  HYPERBILIRUBINEMIA : Total | 1 | 0 | 0 | 1
  LEUKOPENIA : Mild | 1 | 1 | 2 | 1
  LEUKOPENIA : Moderate | 0 | 0 | 0 | 1
  LEUKOPENIA : Severe | 0 | 0 | 0 | 0
  LEUKOPENIA : Total | 1 | 1 | 2 | 2
  NEUTROPENIA : Mild | 1 | 0 | 0 | 1
  NEUTROPENIA : Moderate | 0 | 0 | 0 | 0
  NEUTROPENIA : Severe | 0 | 0 | 0 | 0
  NEUTROPENIA : Total | 1 | 0 | 0 | 1

9. Secondary Outcome: Geometric Mean NiV(M) Pre-F Binding Antibody Titer (GMTs) and 95% Confidence Intervals (CIs).
Description: Vaccine-induced binding antibody titers against Pre-F antigen of Nipah virus Malaysia strain (NiV(M)) were measured by ELISA. The value of the antibody response was determined by obtaining half of the maximum effective concentration (EC50) titer from the optical density 450 nm curves for the function of the reciprocal dilution using a four-parameter logistic curve fit in Prism (version 10.2.2). NiV Pre-F EC50 titers were normalized using the World Health Organization (WHO)/National Institute for Biological Standards and Control (NIBSC) international standard (IS, NIBSC code 22/130) and are reported as group geometric mean titers (GMTs) and 95% confidence intervals (CIs) in international units per milliliter (IU/ml).
Time Frame: Serum samples collected at baseline (Week 0) and at two weeks after the second product administration (Week 6).
Population: Baseline analyses included all study participants who received the first dose (N=40) and Week 6 analyses included all study participants who received both the first and the second doses (N=38). One participant in 10 mcg dose group received only one vaccination and one participant in 25 mcg dose group missed Week 6 visit.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 10 | 10 | 10 | 10
IU/mL
  Week 0 | 4.44 [1.98 to 9.95] | 1.28 [0.83 to 1.97] | 1.83 [1.2 to 2.8] | 3.03 [1.94 to 4.74]
  Week 6: number analyzed (Participants) | 9 | 10 | 10 | 9
  Week 6 | 1941.62 [1168 to 3227.66] | 1885.99 [1025.75 to 3467.66] | 1411.64 [1008.13 to 1976.66] | 923.47 [526.95 to 1618.34]

10. Secondary Outcome: Geometric Mean NiV(M) G Binding Antibody Titer (GMTs) and 95% Confidence Intervals (CIs).
Description: Vaccine-induced binding antibody titers against G antigen of Nipah virus Malaysia strain (NiV(M)) were measured by ELISA. The value of the antibody response was determined by obtaining half of the maximum effective concentration (EC50) titer from the optical density 450 nm curves for the function of the reciprocal dilution using a four-parameter logistic curve fit in Prism (version 10.2.2). NiV G EC50 titers were normalized using the World Health Organization (WHO)/National Institute for Biological Standards and Control (NIBSC) international standard (IS, NIBSC code 22/130) and are reported as group geometric mean titers (GMTs) and 95% confidence intervals (CIs) in international units per milliliter (IU/ml).
Time Frame: Serum samples collected at baseline (Week 0) and at two weeks after the second product administration (Week 6).
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 10 | 10 | 10 | 10
IU/mL
  Week 0 | 12.48 [4.93 to 31.57] | 2.84 [1.72 to 4.68] | 4.12 [2.48 to 6.86] | 6.91 [4.14 to 11.54]
  Week 6: number analyzed (Participants) | 9 | 10 | 10 | 9
  Week 6 | 4626.43 [2962.81 to 7224.18] | 5013 [2717.16 to 9248.69] | 4279.39 [3293.62 to 5560.2] | 2403.1 [1311.35 to 4403.76]

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were reported for 7 days after product administration. Unsolicited AEs were reported for 4 weeks after study product administration. Serious AEs and new chronic medical conditions were reported through last study visit (up to Week 56)
Description: The overall Arms/Groups summarize AEs collected after product administration separately and grouped by the study product and dose. Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment represent the number and percentage of participants reporting the event. A participant with multiple experiences of the same event is counted once using the event of worst severity. Influenza/ILI were collected separately and not included as AE.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 10/10 | 10/10 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=10) | Group 2 (N=10) | Group 3 (N=10) | Group 4 (N=10)
Anemia (Blood and lymphatic system disorders) | 1 | 3 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Injection site bruising (General disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory synctial virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper Respiratory Tract infection (Infections and infestations) | 2 | 1 | 0 | 2
Anthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 2
Malaise (General disorders) | 2 | 6 | 8 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 6 | 2
Headache (Nervous system disorders) | 4 | 4 | 6 | 1
Chills (General disorders) | 1 | 1 | 4 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 1
Pyrexia (General disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 1 — Joint Pain
Administration site pain (General disorders) | 9 | 9 | 9 | 6
Administration site swelling (General disorders) | 0 | 0 | 1 | 0
Administration site erythema (General disorders) | 0 | 0 | 2 | 0
Administration site pruritus (General disorders) | 1 | 0 | 1 | 1
Axillary Lymphadenopathy ipsilateral to the injection site (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-12-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT05398796/Prot_SAP_ICF_001.pdf